CLINICAL TRIAL: NCT07205133
Title: Effectiveness of Whole Body Vibration Therapy and Usual Care Compared to Usual Care in Improving Muscle Mass, Strength and Function in Older Adults
Brief Title: A Randomized Controlled Trial Comparing Whole Body Vibration Therapy With Usual Care and Usual Care to Improve Muscle Health in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Collaborators: BMEC Pte Ltd (Unknown)
Responsible Party: Principal Investigator, Christine Chen Yuanxin, Doctor, Changi General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECOS Ref: 2025-0362; AM/AG001/2025 (SRDUKAMR25G1) (Other Grant/Funding Number: Singhealth Duke-NUS Academic Medicine Research Grant 2.0 FY 2025: Special Category (Ageing Research- AGER))
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Aging; Frailty; Sarcopenia; Muscle Strength; Muscle Function; Muscle Mass
Keywords: Aging; Frailty; Sarcopenia; Whole Body Vibration Therapy; Muscle Strength; Muscle Function; Muscle Mass
MeSH Terms: conditions — Frailty; Sarcopenia

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whole Body Vibration Training (Experimental): The WBVT would be conducted using the Galileo Vibration machine (Galileo® S 35), for 3 sessions per week for 4 weeks.
  The participants would be progressed in terms of (i)vibration frequency from 15 Hz to at least 25 Hz (maximum 30 Hz for those who can tolerate) (ii)for the angles of their squats (from an approximate starting point of 20 degrees ("mini squats" to 45 degrees "quarter squats"; maximum to 90 degrees-thighs parallel to ground or "half-squats" for those who can tolerate); as well as (iii) increasing number of each 1-minute set (from 6 to 8 sets), while standing on the WBVT machine barefoot with both feet flat on the platform set at an amplitude of 2-3mm (according to the participant's height and body physique) with variable rest breaks (up to 1 minute) between each set for a total of 15 minutes each training session.
  Any missed session would be recorded. To ensure compliance, the subjects would receive a standard phone-call/text reminder prior to the scheduled session.
  Interventions: Other: Whole Body Vibration Training; Other: Otago Exercise
- Usual Care (Active Comparator): Participants from both arms would also be provided the exercise sheet on "Otago exercises" (30)and demonstrated in one session how to perform the exercises. In-person demonstration of the "Otago exercises" would be done upon recruitment by trained study team members, at the visit for baseline measurements and a return-demonstration would be done after. They would be instructed to perform the Otago exercises daily according to the standardized instructions stated and progressed from 10 to 15 repetitions on their own for at least 3 times a week and advised to also continue other aerobic exercises, for example, brisk walking. Participants would be given an exercise and falls diary to record their exercise participation as well as any falls that occurred during the study duration for up to 3 months.
  Interventions: Other: Otago Exercise

INTERVENTIONS:
Other: Whole Body Vibration Training — Information already included in arm/group descriptions.
  Arms: Whole Body Vibration Training
Other: Otago Exercise — Usual Care

SUMMARY:
This study is a randomized controlled trial where participants would be randomly assigned to one of 2 groups. One group would receive Whole body vibration therapy and usual care and the other group only usual care. Measurements of muscle mass, strength and function would be taken before the interventions, and at 2 other points after interventions. Differences in the outcomes between the two groups would be analysed.

DETAILED DESCRIPTION:
Background: The prevalence of Frailty and Sarcopenia is increasing with increasing proportion of older adults in the population. While screening for frailty and sarcopenia has become more common, frailty interventions are still developing. Effective interventions include resistance exercise programs that are progressive and sustained. However, take up rate and adherence to these programs are low due to many barriers like time, cost and convenience to the older adult. Many older adults who are frail may be unable to adhere to exercise programs due to cognitive impairment and tolerability. An alternative modality, Whole Body Vibration Training (WBVT), has emerged with evidence in improving muscle strength and function which may be easier to complete and a safe alternative.

Aim: Our study aims to evaluate the effectiveness of a novel progressive 4-week, thrice-weekly WBVT intervention and usual care compared to usual care in improving muscle mass, strength and function in the pre-frail and mildly frail older adult.

Methods: 20 participants would be randomly allocated to each arm. The primary outcome is the between-group difference in change in maximal isometric knee-extension strength from baseline to 2 weeks post-intervention. Secondary outcomes include Appendicular Skeletal Mass Index (ASMI), hand grip strength (HGS), gait speed (GS), 5 timed chair stands, Quality of life (EQ-5D-5L) and physical activity level using the Physical Activity Scale for the Elderly (PASE). Other secondary outcomes include falls rate during the study, 1-year unplanned emergency department visits, hospitalizations as well as all-cause mortality. The measurements would be done at 3 points, namely pre-intervention (baseline), 2 weeks post-intervention and at 3 months. Qualitative data would include participant surveys and semi-structured interviews to assess feasibility, accessibility and future implementation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteer or Patients aged 65 and above,
* Clinical frailty Scale (CFS) score of 3-4,
* Independently ambulating without any aid
* willingness and consent to participate in the study and ability to travel to the study-site for the measurements and interventions, and
* participants with no regular exercise habits (defined as less than 150mins/week of moderate intensity aerobic exercise and less than twice a week of strengthening exercises)for past 3 months.

Exclusion Criteria:

* current active enrolment into any Day Rehab or community exercise program,
* contraindications to WBVT machine usage (see below),
* diagnosis of dementia,
* history of Diabetes Mellitus
* BMI ≤20kg/m2,
* recent hospital admissions within the last 3 months,
* end stage organ failure,
* chronic diseases which are not well managed, for example, poorly controlled hypertension,
* New York Heart Association (NYHA) score II and above for patients with history of heart failure and
* MUST Score ≥1.

Contraindications to WBVT:

PRIMARY CONTRAINDICATIONS TO WBVT

* Pregnancy
* Acute thrombosis (acute vascular occlusion)
* Artificial joints in stimulated body regions
* Fresh fractures in stimulated body regions
* Within 3 months post surgery/procedure and/or any fresh wounds and scars in the stimulated body regions
* or if the wound healing is not yet completely finished.

SECONDARY CONTRAINDICATIONS TO WBVT

* Acute inflammation of the musculoskeletal system, activated arthrosis or
* arthropathy (e.g. acute inflammation and swelling in joints).
* Acute tendinopathies in stimulated body regions (acute tendonitis)
* Acute hernias (tissue ruptures)
* Acute discopathy (acute disc-related back problem)
* Stone disease of the bile ducts and urinary tract
* Rheumatoid Arthritis
* Epilepsy due to secondary risk of injury

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Isometric Knee Extension Strength | Baseline and 2 weeks after intervention and 3 months after intervention
  Measured using a JTech Medical, Northstar Echo Muscle Tester with subject seated with knee flexed at 90 degrees and hanging, muscle tester is placed at the ventral surface of the ankle between malleoli and subject instructed to push against tester with maximal effort to extend the knee. Best of three trials would be taken.

SECONDARY OUTCOMES:
Hand Grip Strength | Baseline and at 2 weeks post intervention and 3 months post intervention
  Measured using Jtech Medical, Northstar Echo Grip hand dynamometer with participant sitting upright with elbows flexed at 90 degrees and arms unsupported, best of 3 tries from each hand.
Appendicular Skeletal Mass Index | Baseline and at 2 weeks post intervention and 3 months post intervention
  Height adjusted Appendicular Skeletal Mass index as measured by the InBody S10 Body Composition Analysis machine
Gait Speed | Baseline and at 2 weeks post intervention and 3 months post intervention
  6 metres normal gait speed (metres/second)
5-timed chair stands | Baseline and at 2 weeks post intervention and 3 months post intervention
  Time taken to perform 5 chair stands with both arms crossed over chest (seconds)
Calf Circumference | Baseline and at 2 weeks post intervention and 3 months post intervention
  Widest calf circumference with participant in standing position
Physical Activity Scale for the Elderly (PASE) | Baseline and at 2 weeks post intervention and 3 months post intervention
  Assessment for physical activity level according to the PASE questionnaire
Quality of life scale | Baseline and at 2 weeks post intervention and 3 months post intervention
  QOL measured with the EQ-5D-5L
Number of falls | 1 year post interventions
  Number of falls per participant during study period
1 year unplanned emergency department visits and hospitalisation events | 1 year post interventions
  as described above
All-cause mortality | up to 1 year post interventions
  Mortality all-cause

OTHER OUTCOMES:
Participant Surveys | 2 weeks post intervention up to 3 months post intervention
  Survey on user experience and satisfaction as well as feasibility, accessibility
Exercise adherence | During 4 weeks intervention period
  Participants would be instructed to record their exercise participation in an exercise diary with remarks on any symptoms experienced.
Semi-structured interviews | 2 weeks post intervention up to 3 months post intervention
  Semi-structured interviews would be conducted for the 20 participants in the WBVT (intervention) arm to enhance the qualitative data collected.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared at this time because participants were not explicitly consented for data sharing.

REFERENCES:
- [Background] Dyer SM, Crotty M, Fairhall N, Magaziner J, Beaupre LA, Cameron ID, Sherrington C; Fragility Fracture Network (FFN) Rehabilitation Research Special Interest Group. A critical review of the long-term disability outcomes following hip fracture. BMC Geriatr. 2016 Sep 2;16(1):158. doi: 10.1186/s12877-016-0332-0. PMID 27590604
- [Background] Akehurst H, Grice JE, Angioi M, Morrissey D, Migliorini F, Maffulli N. Whole-body vibration decreases delayed onset muscle soreness following eccentric exercise in elite hockey players: a randomised controlled trial. J Orthop Surg Res. 2021 Oct 12;16(1):589. doi: 10.1186/s13018-021-02760-4. PMID 34641941
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Lee SY, Goh A, Tan K, Choo PL, Ong PH, Wong WP, Wee SL. Effectiveness of a community-delivered pneumatic machine resistance training programme (Gym Tonic) for older adults at neighbourhood senior centres - a randomized controlled trial. Eur Rev Aging Phys Act. 2021 Oct 7;18(1):21. doi: 10.1186/s11556-021-00273-x. PMID 34620081
- [Background] Claflin DR, Larkin LM, Cederna PS, Horowitz JF, Alexander NB, Cole NM, Galecki AT, Chen S, Nyquist LV, Carlson BM, Faulkner JA, Ashton-Miller JA. Effects of high- and low-velocity resistance training on the contractile properties of skeletal muscle fibers from young and older humans. J Appl Physiol (1985). 2011 Oct;111(4):1021-30. doi: 10.1152/japplphysiol.01119.2010. Epub 2011 Jul 28. PMID 21799130
- [Background] Burd NA, West DW, Staples AW, Atherton PJ, Baker JM, Moore DR, Holwerda AM, Parise G, Rennie MJ, Baker SK, Phillips SM. Low-load high volume resistance exercise stimulates muscle protein synthesis more than high-load low volume resistance exercise in young men. PLoS One. 2010 Aug 9;5(8):e12033. doi: 10.1371/journal.pone.0012033. PMID 20711498
- [Background] Yoshiko A, Watanabe K. Author Correction: Impact of home-based squat training with two-depths on lower limb muscle parameters and physical functional tests in older adults. Sci Rep. 2021 Jul 29;11(1):15802. doi: 10.1038/s41598-021-95096-2. No abstract available. PMID 34326445
- [Background] Chew STH, Kayambu G, Lew CCH, Ng TP, Ong F, Tan J, Tan NC, Tham SL. Singapore multidisciplinary consensus recommendations on muscle health in older adults: assessment and multimodal targeted intervention across the continuum of care. BMC Geriatr. 2021 May 17;21(1):314. doi: 10.1186/s12877-021-02240-8. PMID 34001023
- [Background] Currier BS, Mcleod JC, Banfield L, Beyene J, Welton NJ, D'Souza AC, Keogh JAJ, Lin L, Coletta G, Yang A, Colenso-Semple L, Lau KJ, Verboom A, Phillips SM. Resistance training prescription for muscle strength and hypertrophy in healthy adults: a systematic review and Bayesian network meta-analysis. Br J Sports Med. 2023 Sep;57(18):1211-1220. doi: 10.1136/bjsports-2023-106807. Epub 2023 Jul 6. PMID 37414459
- [Background] Hurst C, Robinson SM, Witham MD, Dodds RM, Granic A, Buckland C, De Biase S, Finnegan S, Rochester L, Skelton DA, Sayer AA. Resistance exercise as a treatment for sarcopenia: prescription and delivery. Age Ageing. 2022 Feb 2;51(2):afac003. doi: 10.1093/ageing/afac003. PMID 35150587
- [Background] Wu S, Ning HT, Xiao SM, Hu MY, Wu XY, Deng HW, Feng H. Effects of vibration therapy on muscle mass, muscle strength and physical function in older adults with sarcopenia: a systematic review and meta-analysis. Eur Rev Aging Phys Act. 2020 Sep 17;17:14. doi: 10.1186/s11556-020-00247-5. eCollection 2020. PMID 32963629
- [Background] Yi M, Zhang W, Zhang X, Zhou J, Wang Z. The effectiveness of Otago exercise program in older adults with frailty or pre-frailty: A systematic review and meta-analysis. Arch Gerontol Geriatr. 2023 Nov;114:105083. doi: 10.1016/j.archger.2023.105083. Epub 2023 Jun 22. PMID 37390692
- [Background] Lam FM, Lau RW, Chung RC, Pang MY. The effect of whole body vibration on balance, mobility and falls in older adults: a systematic review and meta-analysis. Maturitas. 2012 Jul;72(3):206-13. doi: 10.1016/j.maturitas.2012.04.009. Epub 2012 May 18. PMID 22609157
- [Background] Remer F, Keilani M, Kull P, Crevenna R. Effects of whole-body vibration therapy on pain, functionality, postural stability, and proprioception in patients with subacute and chronic non-specific low back pain: a systematic review. Wien Med Wochenschr. 2025 Feb;175(1-2):20-40. doi: 10.1007/s10354-023-01026-4. Epub 2023 Nov 24. PMID 37999785
- [Background] Gloeckl R, Heinzelmann I, Kenn K. Whole body vibration training in patients with COPD: A systematic review. Chron Respir Dis. 2015 Aug;12(3):212-21. doi: 10.1177/1479972315583049. Epub 2015 Apr 22. PMID 25904085
- [Background] Nowak-Lis A, Nowak Z, Gabrys T, Szmatlan-Gabrys U, Batalik L, Knappova V. The Use of Vibration Training in Men after Myocardial Infarction. Int J Environ Res Public Health. 2022 Mar 11;19(6):3326. doi: 10.3390/ijerph19063326. PMID 35329010
- [Background] Qiu CG, Chui CS, Chow SKH, Cheung WH, Wong RMY. Effects of Whole-Body Vibration Therapy on Knee Osteoarthritis: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Rehabil Med. 2022 Mar 29;54:jrm00266. doi: 10.2340/jrm.v54.2032. PMID 35174868
- [Background] Yang X, Xue X, Tu H, Li N. Effect of whole-body vibration training on the recovery of lower limb function in people with stroke: a systematic review and meta-analysis. Disabil Rehabil. 2023 Nov;45(23):3823-3832. doi: 10.1080/09638288.2022.2138993. Epub 2022 Nov 11. PMID 36367314
- [Background] Costantino C, Bertuletti S, Romiti D. Efficacy of Whole-Body Vibration Board Training on Strength in Athletes After Anterior Cruciate Ligament Reconstruction: A Randomized Controlled Study. Clin J Sport Med. 2018 Jul;28(4):339-349. doi: 10.1097/JSM.0000000000000466. PMID 28657911
- [Background] Lai CC, Tu YK, Wang TG, Huang YT, Chien KL. Effects of resistance training, endurance training and whole-body vibration on lean body mass, muscle strength and physical performance in older people: a systematic review and network meta-analysis. Age Ageing. 2018 May 1;47(3):367-373. doi: 10.1093/ageing/afy009. PMID 29471456
- [Background] Billot M, Calvani R, Urtamo A, Sanchez-Sanchez JL, Ciccolari-Micaldi C, Chang M, Roller-Wirnsberger R, Wirnsberger G, Sinclair A, Vaquero-Pinto N, Jyvakorpi S, Ohman H, Strandberg T, Schols JMGA, Schols AMWJ, Smeets N, Topinkova E, Michalkova H, Bonfigli AR, Lattanzio F, Rodriguez-Manas L, Coelho-Junior H, Broccatelli M, D'Elia ME, Biscotti D, Marzetti E, Freiberger E. Preserving Mobility in Older Adults with Physical Frailty and Sarcopenia: Opportunities, Challenges, and Recommendations for Physical Activity Interventions. Clin Interv Aging. 2020 Sep 16;15:1675-1690. doi: 10.2147/CIA.S253535. eCollection 2020. PMID 32982201
- [Background] Ng TP, Feng L, Nyunt MS, Feng L, Niti M, Tan BY, Chan G, Khoo SA, Chan SM, Yap P, Yap KB. Nutritional, Physical, Cognitive, and Combination Interventions and Frailty Reversal Among Older Adults: A Randomized Controlled Trial. Am J Med. 2015 Nov;128(11):1225-1236.e1. doi: 10.1016/j.amjmed.2015.06.017. Epub 2015 Jul 6. PMID 26159634
- [Background] Lim WS, Cheong CY, Lim JP, Tan MMY, Chia JQ, Malik NA, Tay L. Singapore Clinical Practice Guidelines For Sarcopenia: Screening, Diagnosis, Management and Prevention. J Frailty Aging. 2022;11(4):348-369. doi: 10.14283/jfa.2022.59. PMID 36346721
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Dent E, Lien C, Lim WS, Wong WC, Wong CH, Ng TP, Woo J, Dong B, de la Vega S, Hua Poi PJ, Kamaruzzaman SBB, Won C, Chen LK, Rockwood K, Arai H, Rodriguez-Manas L, Cao L, Cesari M, Chan P, Leung E, Landi F, Fried LP, Morley JE, Vellas B, Flicker L. The Asia-Pacific Clinical Practice Guidelines for the Management of Frailty. J Am Med Dir Assoc. 2017 Jul 1;18(7):564-575. doi: 10.1016/j.jamda.2017.04.018. PMID 28648901
- [Background] Dent E, Martin FC, Bergman H, Woo J, Romero-Ortuno R, Walston JD. Management of frailty: opportunities, challenges, and future directions. Lancet. 2019 Oct 12;394(10206):1376-1386. doi: 10.1016/S0140-6736(19)31785-4. PMID 31609229
- [Background] Dent E, Chapman I, Howell S, Piantadosi C, Visvanathan R. Frailty and functional decline indices predict poor outcomes in hospitalised older people. Age Ageing. 2014 Jul;43(4):477-84. doi: 10.1093/ageing/aft181. Epub 2013 Nov 19. PMID 24257468
- [Background] Hoogendijk EO, Afilalo J, Ensrud KE, Kowal P, Onder G, Fried LP. Frailty: implications for clinical practice and public health. Lancet. 2019 Oct 12;394(10206):1365-1375. doi: 10.1016/S0140-6736(19)31786-6. PMID 31609228
- See also: Ministry of Health Singapore. MOH Frailty Strategy Policy Report [Internet]. [cited 2024 Sep 5] — https://www.moh.gov.sg/resources-statistics/reports/frailty-strategy-policy-report
- See also: Ministry of Health Singapore. National Population Healthy Survey 2022 [Internet]. [cited 2024 Sep 5] — https://www.moh.gov.sg/resources-statistics/reports/national-population-health-survey-2022
- See also: Ministry of Health Singapore. The White Paper on Healthier SG [Internet]. [cited 2024 Sep 5] — https://www.healthiersg.gov.sg/resources/white-paper/